CLINICAL TRIAL: NCT04405960
Title: Role of Vitamin D (Alphacalcidol) Supplement to Reduce Pain and Cartilage Oligomeric Matrix Protein Serum Levels in Geriatric Knee Osteoarthritis Patients: A Randomized, Double-Blind, Placebo-Controlled Study
Brief Title: Role of Alphacalcidol Supplement to Reduce Pain and COMP in Geriatric Knee Osteoarthritis Patients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Syarif Hidayatullah State Islamic University Jakarta (Other)
Responsible Party: Principal Investigator, Achmad Zaki, Doctor, Orthopedic Surgeon, Principal Investigator, Syarif Hidayatullah State Islamic University Jakarta
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 162/UN2.F10/PPM.00.02/2016
Record Dates: First submitted 2020-05-14; First posted 2020-05-28 (Actual); Last update posted 2020-05-28 (Actual); Status verified 2020-05

CONDITIONS: Osteoarthritis, Knee; Aged
Keywords: Vitamin D; Alfacalcidol; Knee osteoarthritis pain; Cartilage Oligomeric Matrix Protein
MeSH Terms: conditions — Osteoarthritis, Knee; Pseudoachondroplasia | interventions — alfacalcidol; Sugars

STUDY DESIGN:
Intervention Model Description: This is a randomized, double-blind, and placebo-controlled trials. Elderly subjects with symptomatic knee OA visited our clinic in Jakarta were recruited. Medical history taking, physical examinations, knee radiology, blood test for Vitamin D (25(OH)D), calcium, and COMP serum were performed. Subjects were then randomly allocated to either intervention group to be given 1 µg Alphacalcidol or control group to be given placebo in 12 weeks.
Who Masked: Participant, Care Provider, Investigator
Masking Description: This study used Contract Research Organization (CRO) Equilab to ensure the quality. In this study, researchers, respondents, interviewers, supplement providers, radiology and laboratory staffs were blinded. The interviewers used a questionnaire that had been prepared previously and was used equally for the intervention and control groups.
  Knee x-ray examination was performed to determine knee OA severity based on Kellgren-Lawrence grading system. It was carried out using the same method and technique between the intervention and control groups. X-ray examination was carried out at the same hospital's radiology unit and was interpreted blindingly by the same radiologist. Blood examination to measure 25(OH)D and COMP was carried out using the same methods and techniques between the intervention and control groups by staffs from the same certified laboratory.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): Individuals in intervention group were given oral Vitamin D supplements (Alphacalcidol 1 µg) once daily
  Interventions: Drug: Alfacalcidol 1 MCG Oral Capsule
- Control Group (Placebo Comparator): Individuals in control group were given placebo once daily
  Interventions: Drug: Sugar pill

INTERVENTIONS:
Drug: Alfacalcidol 1 MCG Oral Capsule — The subjects in the intervention group were given 1 µg oral capsule alphacalcidol once daily Subjects in the control group were given placebo once daily with similar capsule shape and color to the capsule given to the intervention group. The process of alphacalcidol and placebo encapsulation were carried out by pharmacists in the pharmacy depot under the supervision of researchers and CRO Equilab. Alphacalcidol and placebo were put into plastic pots containing 30 capsules for every 4 weeks for each subject. The pot had an etiquette written explaining how to consume the drug (after breakfast between 7 - 10 a.m.). The drugs' packaging and code numbering were carried out by CRO Equilab to ensure a double-blind procedure. As a control, each subject was equipped with a monitoring card. Alphacalcidol and placebo were given for 12 weeks without interruption. Monitoring of compliance and side effects was performed by physicians every 2 weeks.
  Other Names: Bon-One; One-Alpha
  Arms: Intervention group
Drug: Sugar pill — The subjects in the control group were given placebo containing simple sugar oral capsule once daily with similar capsule shape and color to the capsule given to the intervention group. The process of alphacalcidol and placebo encapsulation were carried out by pharmacists in the pharmacy depot under the supervision of researchers and CRO Equilab. Alphacalcidol and placebo were put into plastic pots containing 30 capsules for every 4 weeks for each subject. The pot had an etiquette written explaining how to consume the drug (after breakfast between 7 - 10 a.m.). The drugs' packaging and code numbering were carried out by CRO Equilab to ensure a double-blind procedure. As a control, each subject was equipped with a monitoring card. Alphacalcidol and placebo were given for 12 weeks without interruption. Monitoring of compliance and side effects was performed by physicians every 2 weeks.
  Other Names: Placebo
  Arms: Control Group

SUMMARY:
Indonesian population's life expectancy has been increasing steadily in the last 3 decades. It potentially increases the prevalence of degenerative diseases, including osteoarthritis (OA). Serum Vitamin D (25(OH)D) level has been recognized as a risk factors for knee OA. Cartilage Oligomeric Matrix Protein (COMP) is cartilage degradation product can be used as a diagnostic marker for knee OA. This study aims to determine the effect of Vitamin D supplementation (Alphacalcidol) on pain based on WOMAC indicators and joint cartilage condition based on COMP serum markers in knee OA elderly patients.

DETAILED DESCRIPTION:
Vitamin D plays important role to enhance calcium absorption in intestine and promotes mineralization of bones. Several studies found that Vitamin D levels were low in patients with knee OA.

Vitamin D deficiency were found in 50% of women age 45-55 years old and 35% of women age 60-90 years old in Jakarta and Bekasi. Alphacalcidol is a vitamin D supplementation recommended to be used in patients with renal insufficiency, which is prevalent in elderly. Alfacalcidol does not need to undergo renal 1-alpha-hydroxylation which impaired in renal insufficiency, although it can still cause hypercalcemia.

Current detection and diagnosis of knee OA relies on plain radiological examination, which is not really objective because it depends on radiological expertise and experience. Moreover, plain radiological diagnosis has limited ability to detect joint damage at an early stage. Therefore, knee OA is often diagnosed at advanced stage. For this reason, selecting accurate joint cartilage biomarkers is important to detect and predict the severity of OA objectively and at earlier stage. Cartilage Oligomeric Matrix Protein (COMP) is one of degradation products released into synovium fluid and bloodstream from cartilage matrix turnover process. Therefore, COMP can be used as a marker of diagnosis and cartilage injury severity of knee OA.

Currently, there has been no study about the association of Vitamin D supplementation with pain level and cartilage matrix turnover process in Indonesia. Therefore, this study aims to determine the effect of Vitamin D supplementation (Alphacalcidol) on pain and joint cartilage condition in elderly patients with knee OA.

ELIGIBILITY:
Inclusion Criteria:

* Patients with knee pain due to OA who meet clinical and radiological criteria according to Kellgren-Lawrence grade at least 1 month with knee pain of at least 5 measured using the WOMAC pain index
* Body mass index ≤27 kg/m2
* Do not have any systemic inflammatory diseases or other systemic diseases from history taking and physical examination
* Do not have any other OA in other joints according to physical examination
* Did not do any heavy physical activity or strenuous exercise for at least 1 month (last month)

Exclusion Criteria:

* Grade 4 Kellgren-Lawrence
* WOMAC pain score >15
* Serum 25(OH)D >125 nmol/L
* Calcium serum >10.5 mg/dl
* Diagnosed with rheumatoid or psoriatic arthritis, lupus or cancer, heart or kidney disorders, vitamin D hypersensitivity.
* Knee trauma, including injury to the ligament or meniscus before the study
* Consuming drugs that contain Magnesium (Antacids), Digitalis (Digoxin), Barbiturates or other anti-convulsants for a long time, which will interact with Vitamin D
* Currently undergoing vitamin D therapy for the last 30 days
* Use of other supplements intended to have an effect on cartilage such as glucosamine and chondroitin sulphate
* Undergo intra-articular therapy 3 months before the study
* Consume oral corticosteroids
* Senile dementia or other signs and symptoms of memory loss

Ages: 60 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 146 (Actual)
Dates: Start 2017-07-01 (Actual); Primary Completion 2017-09-30 (Actual); Study Completion 2017-12-31 (Actual)

PRIMARY OUTCOMES:
WOMAC Pain Score Difference | Initial and final week (week 0 and 12).
  Instrument for assessing pain in knee OA patients from The Western Ontario & McMaster University OA Index. WOMAC pain score was assessed every 2 weeks to ensure that subject's pain within inclusion criteria.
Cartilage Oligomeric Matrix Protein Difference | Initial and final week (week 0 and 12).
  Serum concentration of Cartilage Oligomeric Matrix Protein (COMP) as a biomarker for the severity of knee OA.

SECONDARY OUTCOMES:
Serum 25(OH)D Concentration Difference | Initial and final week (week 0 and 12).
  Serum 25(OH)D Concentration as vitamin D deficiency status
Body Mass Index | Once, on week-0
  Body mass index, calculated by measuring subject's height and weight
Kellgren-Lawrence Knee OA Grade | Once, on week-0
  Radiological knee OA grading system
Mean Physical Activity | Every 2 weeks (from week-0 until week-12)
  Physical activities performed by subjects using their energy related to work and daily leisure time. Measured using Basic Health Research (Riskesdas) 2007 Questionnaire
Mean Sun Exposure Frequency | Every 2 weeks (from week-0 until week-12)
  Ultraviolet B (UVB) exposure between 7-11 am for ≥ 30 minutes with exposure at least to the face and palms
Mean Vitamin D Consumption | Every 4 weeks (from week-0 until week-12)
  The amount of Vitamin D consumption by subjects, which is calculated based on the consumption of fruits, vegetables, milk and its processed products, fish, etc.

CONTACTS AND LOCATIONS:
Overall Officials: Achmad Zaki, PhD, Principal Investigator — Faculty of Medicine Syarif Hidayatullah State Islamic University Jakarta
Locations (1):
- Public Health Service Clinic Reni Jaya, South Tangerang, Banten, Indonesia

IPD SHARING:
Plan to Share IPD: No
Author's informed consent does not include IPD sharing agreement.

REFERENCES:
- [Background] Gueli N, Verrusio W, Linguanti A, Di Maio F, Martinez A, Marigliano B, Cacciafesta M. Vitamin D: drug of the future. A new therapeutic approach. Arch Gerontol Geriatr. 2012 Jan-Feb;54(1):222-7. doi: 10.1016/j.archger.2011.03.001. Epub 2011 Apr 1. PMID 21458871
- [Background] Bassiouni H, Aly H, Zaky K, Abaza N, Bardin T. Probing The Relation Between Vitamin D Deficiency and Progression of Medial Femoro-tibial Osteoarthitis of the Knee. Curr Rheumatol Rev. 2017;13(1):65-71. doi: 10.2174/1573397112666160404124532. PMID 27041085
- [Background] Veronese N, Maggi S, Noale M, De Rui M, Bolzetta F, Zambon S, Corti MC, Sartori L, Musacchio E, Baggio G, Perissinotto E, Crepaldi G, Manzato E, Sergi G. Serum 25-Hydroxyvitamin D and Osteoarthritis in Older People: The Progetto Veneto Anziani Study. Rejuvenation Res. 2015 Dec;18(6):543-53. doi: 10.1089/rej.2015.1671. Epub 2015 Nov 5. PMID 26540555
- [Background] Jansen JA, Haddad FS. High prevalence of vitamin D deficiency in elderly patients with advanced osteoarthritis scheduled for total knee replacement associated with poorer preoperative functional state. Ann R Coll Surg Engl. 2013 Nov;95(8):569-72. doi: 10.1308/rcsann.2013.95.8.569. PMID 24165338
- [Background] Oemardi M, Horowitz M, Wishart JM, Morris HA, Need AG, O'loughlin PD, Nordin BE. The effect of menopause on bone mineral density and bone-related biochemical variables in Indonesian women. Clin Endocrinol (Oxf). 2007 Jul;67(1):93-100. doi: 10.1111/j.1365-2265.2007.02844.x. Epub 2007 May 9. PMID 17490404
- [Background] Ebeling PR, Adler RA, Jones G, Liberman UA, Mazziotti G, Minisola S, Munns CF, Napoli N, Pittas AG, Giustina A, Bilezikian JP, Rizzoli R. MANAGEMENT OF ENDOCRINE DISEASE: Therapeutics of Vitamin D. Eur J Endocrinol. 2018 Oct 12;179(5):R239-R259. doi: 10.1530/EJE-18-0151. PMID 30131372
- [Background] Palmer SC, McGregor DO, Craig JC, Elder G, Macaskill P, Strippoli GF. Vitamin D compounds for people with chronic kidney disease requiring dialysis. Cochrane Database Syst Rev. 2009 Oct 7;(4):CD005633. doi: 10.1002/14651858.CD005633.pub2. PMID 19821349
- [Background] Bartels EM, Christensen R, Christensen P, Henriksen M, Bennett A, Gudbergsen H, Boesen M, Bliddal H. Effect of a 16 weeks weight loss program on osteoarthritis biomarkers in obese patients with knee osteoarthritis: a prospective cohort study. Osteoarthritis Cartilage. 2014 Nov;22(11):1817-25. doi: 10.1016/j.joca.2014.07.027. Epub 2014 Aug 12. PMID 25106676
- [Background] Verma P, Dalal K. Serum cartilage oligomeric matrix protein (COMP) in knee osteoarthritis: a novel diagnostic and prognostic biomarker. J Orthop Res. 2013 Jul;31(7):999-1006. doi: 10.1002/jor.22324. Epub 2013 Feb 19. PMID 23423905
- [Background] Dirks NF, Ackermans MT, Lips P, de Jongh RT, Vervloet MG, de Jonge R, Heijboer AC. The When, What & How of Measuring Vitamin D Metabolism in Clinical Medicine. Nutrients. 2018 Apr 13;10(4):482. doi: 10.3390/nu10040482. PMID 29652819
- [Background] Holick MF. Vitamin D status: measurement, interpretation, and clinical application. Ann Epidemiol. 2009 Feb;19(2):73-8. doi: 10.1016/j.annepidem.2007.12.001. Epub 2008 Mar 10. PMID 18329892
- [Background] Holick MF. High prevalence of vitamin D inadequacy and implications for health. Mayo Clin Proc. 2006 Mar;81(3):353-73. doi: 10.4065/81.3.353. PMID 16529140
- [Background] Ross AC, Manson JE, Abrams SA, Aloia JF, Brannon PM, Clinton SK, Durazo-Arvizu RA, Gallagher JC, Gallo RL, Jones G, Kovacs CS, Mayne ST, Rosen CJ, Shapses SA. The 2011 report on dietary reference intakes for calcium and vitamin D from the Institute of Medicine: what clinicians need to know. J Clin Endocrinol Metab. 2011 Jan;96(1):53-8. doi: 10.1210/jc.2010-2704. Epub 2010 Nov 29. PMID 21118827
- [Background] KELLGREN JH, LAWRENCE JS. Radiological assessment of osteo-arthrosis. Ann Rheum Dis. 1957 Dec;16(4):494-502. doi: 10.1136/ard.16.4.494. No abstract available. PMID 13498604
- [Background] Guermazi A, Hayashi D, Roemer F, Felson DT, Wang K, Lynch J, Amin S, Torner J, Lewis CE, Nevitt MC. Severe radiographic knee osteoarthritis--does Kellgren and Lawrence grade 4 represent end stage disease?--the MOST study. Osteoarthritis Cartilage. 2015 Sep;23(9):1499-505. doi: 10.1016/j.joca.2015.04.018. Epub 2015 Apr 28. PMID 25929973
- [Background] Katz JN, Earp BE, Gomoll AH. Surgical management of osteoarthritis. Arthritis Care Res (Hoboken). 2010 Sep;62(9):1220-8. doi: 10.1002/acr.20231. No abstract available. PMID 20506552
- [Background] Chapple CM, Nicholson H, Baxter GD, Abbott JH. Patient characteristics that predict progression of knee osteoarthritis: a systematic review of prognostic studies. Arthritis Care Res (Hoboken). 2011 Aug;63(8):1115-25. doi: 10.1002/acr.20492. PMID 21560257
- [Background] Jin X, Jones G, Cicuttini F, Wluka A, Zhu Z, Han W, Antony B, Wang X, Winzenberg T, Blizzard L, Ding C. Effect of Vitamin D Supplementation on Tibial Cartilage Volume and Knee Pain Among Patients With Symptomatic Knee Osteoarthritis: A Randomized Clinical Trial. JAMA. 2016 Mar 8;315(10):1005-13. doi: 10.1001/jama.2016.1961. PMID 26954409
- [Background] Ringe JD, Faber H, Fahramand P, Schacht E. Alfacalcidol versus plain vitamin D in the treatment of glucocorticoid/inflammation-induced osteoporosis. J Rheumatol Suppl. 2005 Sep;76:33-40. PMID 16142849
- [Background] Schlogl M, Chocano-Bedoya P, Dawson-Hughes B, Orav EJ, Freystaetter G, Theiler R, Kressig RW, Egli A, Bischoff-Ferrari HA. Effect of Monthly Vitamin D on Chronic Pain Among Community-Dwelling Seniors: A Randomized, Double-Blind Controlled Trial. J Am Med Dir Assoc. 2019 Mar;20(3):356-361. doi: 10.1016/j.jamda.2018.09.004. Epub 2018 Nov 3. PMID 30401610
- [Background] Muraki S, Dennison E, Jameson K, Boucher BJ, Akune T, Yoshimura N, Judge A, Arden NK, Javaid K, Cooper C. Association of vitamin D status with knee pain and radiographic knee osteoarthritis. Osteoarthritis Cartilage. 2011 Nov;19(11):1301-6. doi: 10.1016/j.joca.2011.07.017. Epub 2011 Aug 16. PMID 21884812
- [Background] Bennell KL, Hunter DJ, Hinman RS. Management of osteoarthritis of the knee. BMJ. 2012 Jul 30;345:e4934. doi: 10.1136/bmj.e4934. No abstract available. PMID 22846469
- [Background] Muraki S, Oka H, Akune T, Mabuchi A, En-yo Y, Yoshida M, Saika A, Suzuki T, Yoshida H, Ishibashi H, Yamamoto S, Nakamura K, Kawaguchi H, Yoshimura N. Prevalence of radiographic knee osteoarthritis and its association with knee pain in the elderly of Japanese population-based cohorts: the ROAD study. Osteoarthritis Cartilage. 2009 Sep;17(9):1137-43. doi: 10.1016/j.joca.2009.04.005. Epub 2009 Apr 17. PMID 19410032
- [Background] Vanlint S. Vitamin D and obesity. Nutrients. 2013 Mar 20;5(3):949-56. doi: 10.3390/nu5030949. PMID 23519290
- [Background] Salehpour A, Hosseinpanah F, Shidfar F, Vafa M, Razaghi M, Dehghani S, Hoshiarrad A, Gohari M. A 12-week double-blind randomized clinical trial of vitamin D(3) supplementation on body fat mass in healthy overweight and obese women. Nutr J. 2012 Sep 22;11:78. doi: 10.1186/1475-2891-11-78. PMID 22998754
- [Background] Andersen RE, Crespo CJ, Ling SM, Bathon JM, Bartlett SJ. Prevalence of significant knee pain among older Americans: results from the Third National Health and Nutrition Examination Survey. J Am Geriatr Soc. 1999 Dec;47(12):1435-8. doi: 10.1111/j.1532-5415.1999.tb01563.x. PMID 10591238
- [Background] Ding C, Cicuttini F, Parameswaran V, Burgess J, Quinn S, Jones G. Serum levels of vitamin D, sunlight exposure, and knee cartilage loss in older adults: the Tasmanian older adult cohort study. Arthritis Rheum. 2009 May;60(5):1381-9. doi: 10.1002/art.24486. PMID 19404958
- [Background] Jungert A, Spinneker A, Nagel A, Neuhauser-Berthold M. Dietary intake and main food sources of vitamin D as a function of age, sex, vitamin D status, body composition, and income in an elderly German cohort. Food Nutr Res. 2014 Sep 17;58. doi: 10.3402/fnr.v58.23632. eCollection 2014. PMID 25317118
- [Background] Sanghi D, Mishra A, Sharma AC, Singh A, Natu SM, Agarwal S, Srivastava RN. Does vitamin D improve osteoarthritis of the knee: a randomized controlled pilot trial. Clin Orthop Relat Res. 2013 Nov;471(11):3556-62. doi: 10.1007/s11999-013-3201-6. Epub 2013 Aug 1. PMID 23904246
- [Background] Wu Z, Malihi Z, Stewart AW, Lawes CM, Scragg R. Effect of Vitamin D Supplementation on Pain: A Systematic Review and Meta-analysis. Pain Physician. 2016 Sep-Oct;19(7):415-27. PMID 27676659
- [Background] Corvol MT, Dumontier MF, Tsagris L, Lang F, Bourguignon J. [Cartilage and vitamin D in vitro (author's transl)]. Ann Endocrinol (Paris). 1981 Oct-Nov;42(4-5):482-7. French. PMID 6280580
- [Background] Wislowska M, Jablonska B. Serum cartilage oligomeric matrix protein (COMP) in rheumatoid arthritis and knee osteoarthritis. Clin Rheumatol. 2005 Jun;24(3):278-84. doi: 10.1007/s10067-004-1000-x. Epub 2004 Nov 18. PMID 15940561
- [Background] Clark AG, Jordan JM, Vilim V, Renner JB, Dragomir AD, Luta G, Kraus VB. Serum cartilage oligomeric matrix protein reflects osteoarthritis presence and severity: the Johnston County Osteoarthritis Project. Arthritis Rheum. 1999 Nov;42(11):2356-64. doi: 10.1002/1529-0131(199911)42:113.0.CO;2-R. PMID 10555031
- [Background] Andersson ML, Thorstensson CA, Roos EM, Petersson IF, Heinegard D, Saxne T. Serum levels of cartilage oligomeric matrix protein (COMP) increase temporarily after physical exercise in patients with knee osteoarthritis. BMC Musculoskelet Disord. 2006 Dec 7;7:98. doi: 10.1186/1471-2474-7-98. PMID 17156423